CLINICAL TRIAL: NCT04084834
Title: Feasibility of a Web-based, Peer-supported Exercise Program for Patients With Hip and/or Knee Osteoarthritis
Acronym: AktiWeb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: The Norwegian Rheumatism Association (Other); University of Melbourne (Other); Extrastiftelsen (Other)
Responsible Party: Principal Investigator, Anne Therese Tveter, Physiotherapist, PhD, Diakonhjemmet Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/2198-feasibility
Record Dates: First submitted 2019-08-21; First posted 2019-09-10 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A pre-post single arm feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants allocated to the intervention group will be familiarized with exercise intensity levels (heart rate and Borg RPE) during the assessment at Diakonhjemmet Hospital. Further, the patients will be offered to take part in a 5-hour Learning and Mastery-course at Diakonhjemmet Hospital. Thereafter, the participants will get access to a web-based exercise program and guided to choose the appropriate exercise-level. Weekly, based on the individual progression, all participants will receive an exercise program by email consisting of individually tailored exercise sessions and motivational messages. At the end of each week, the participants complete an electronic exercise diary for monitoring adherence. All participants will be offered the possibility to seek peer-support; however, if preferred they may also follow the exercise program by themselves.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will be offered to take part in a 5-hour Learning and Mastery-course at Diakonhjemmet Hospital, receiving information about the osteoarthritis disease, symptoms and the importance of exercise and physical activity. Participants will then be given a weekly web-based exercise program (12 weeks) consisting of three aerobic exercise sessions per week. The exercise program consists of five levels, and the participants will each week be guided to the most appropriate level based on their measured physical fitness level and the weekly exercise diary. The participants will at initial assessment at Diakonhjemmet Hospital be instructed to use Borgs scale to adjust exercise level. Based on the weekly exercise diary the participants will also get motivational messages by email.

SUMMARY:
In this project, a web-based exercise program is developed in co-creation between specialized health care, the Norwegian Association for Rheumatic diseases (NRF) and a group of experienced patient representatives. The project emerges from the evidence that exercise is recommended as first-line treatment for patients with chronic diseases like hip- and knee-osteoarthritis (OA). However, the number of patients in need of targeted exercise will increase considerably the next decades, and their treatment needs cannot be fully handled within the health care system. Development of innovative and effective treatment trajectories and follow-up strategies is urgently required. Peer-support is recognized as an effective way to increase patients' long-term adherence to exercise. Thus, patient-organizations may be an unutilized resource in support and follow-up of patients who need long-term exercise as part of their treatment plan. After discharge from examination in hospital, patients with hip/knee OA will be recruited to follow-up in a novel web-based, peer-supported exercise program, and the feasibility of the intervention will be evaluated.

DETAILED DESCRIPTION:
The study will be conducted as a pre-post single-arm feasibility study comprising 50 participants.

The main objective of the study will be to evaluate the feasibility of the web-based, peer-supported exercise intervention in patients with hip and/or knee OA.

Specific research objectives are:

* to assess feasibility of intervention delivery, data collection, eligibility and inclusion/exclusion criteria and intervention fidelity
* to assess the responsiveness of relevant primary and secondary outcome measures

In the feasibility study, all participants will be allocated to an intervention group, receiving a 12-week web-based, peer-supported aerobic exercise program including weekly motivational messages. Patients between 40 and 80 years of age that are not candidates for surgery will be recruited from Diakonhjemmet Hospital, Oslo, Norway.

To assess and evaluate feasibility, we will report on descriptive statistics. Responsiveness will be assessed using Receiver Operating Curve (ROC) analyses.

ELIGIBILITY:
Inclusion Criteria:

• patients with hip and/or knee osteoarthritis being referred to Diakonhjemmet Hospital

Exclusion Criteria:

* candidate for surgery
* unable to understand or write Norwegian
* unable to walk unaided and continuously for 15 minutes
* absolute or relative contradictions to maximal exercise testing
* have relatives with sudden death before 40 years of age
* have first-degree relatives with hypertrophic cardiomyopathy

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female gender is a predictor of osteoarthritis, so we expect that more women will be eligible
Enrollment: 31 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility: time resources used by peer-supporters | baseline to 12 weeks
  Time (hours/minutes) per participant-peer-support contact (frequency of contacts divided by total time used by peer-supporters).
Feasibility: time resources used on the exercise program delivery | baseline to 12 weeks
  Time (hours/minutes) per week per participant used on web-based exercise program delivery.
Feasibility: time resources used on motivational messages delivery | baseline to 12 weeks
  Time (hours/minutes) per week per participant used on motivational message delivery.
Feasibility: proportion of received exercise diaries | baseline to 12 weeks
  Proportion of received exercise diaries (0-12 per participant).
Feasibility: proportion wearing the activity monitor | baseline
  Proportion of participants providing activity monitor data (at least 4 days, including one weekend day, with minimum 10 hours recording per day) at baseline.
Feasibility: proportion completing treadmill test | baseline
  Proportion of participants completing the indirect maximal cardiorespiratory exercise test according to test-protocol at baseline.
Eligible: proportion eligible | baseline
  Proportion of potentially eligible participants approached that are invited.
Recruitment: proportion enrolled | baseline
  Proportion of eligible patients enrolled.
Retention: proportion of enrolled participants | baseline and 12 weeks
  Proportion of enrolled participants providing data at 12 week post-test.
Adverse events: number of adverse events | 12 weeks
  Total number of adverse events (by cause if possible) evaluated by answers at post-test: The four questions addressing possible adverse events: 1) Have you carried out any type of treatment during the last 3 months? (With treatment we mean medication, physical exercise, self-management course or any alternative treatments) (yes/no), 2) If yes, have you experienced any adverse event as a result of the treatment? (yes/no). 3) If yes, which adverse events as a result of treatment? 4) In your opinion, which treatment(s) do you think the adverse event was/were caused by? (medication, physical exercise, self-management course, alternative treatments, other) (Elaborate).

SECONDARY OUTCOMES:
Changes in objectively measured physical activity | baseline and 12 weeks
  Assessed by accelerometer (ActiGraph GT3X+): Change in physical activity level measured as counts per minute (CPM), which is the total number of registered counts for all valid days divided by wear time. Thresholds for CPM will be used in calculation of time (minutes per week/day) spent on sitting (<100 CPM), and on light (100-2019 CPM), moderate-(>2019-5998 CPM) and vigorous (>5998) intensity physical activity.
Change in physical fitness (VO2 peak) | baseline and 12 weeks
  Change in VO2 peak measured by indirect maximal cardiorespiratory exercise test (modified Balke-protocol). The indirect estimation of VO2 peak by prediction equations is based on incline, grade and speed at end stage, weight and age.
Change in Hip disability and Osteoarthritis Outcome Score (HOOS) | baseline and 12 weeks
  Change in the last week disability on five subscales; pain (10 items, scale 0-40), symptoms (5 items, scale 0-20), function in daily living (17 items, scale 0-68), function in sport and recreation (4 items, scale 0-16) and quality of life (4 items, scale 0-16). Items are scored by a five-point Likert scale ranging from 0 (least severe) to 4 (most severe). Total sum-score and subscale sum-scores will be converted to normalized scores ranging from 0 (extreme disability) to 100 (no disability).
Change in Knee disability and Osteoarthritis Outcome Score (KOOS) | baseline and 12 weeks
  Change in the last week disability on five subscales; pain (9 items, scale 0-36), symptoms (7 items, scale 0-28), function in daily living (17 items, scale 0-68), function in sport and recreation (5 items, scale 0-20) and quality of life (4 items, scale 0-16). Items are scored by a five-point Likert scale ranging from 0 (least severe) to 4 (most severe). Total sum-score and subscale sum-scores will be converted to normalized scores ranging from 0 (extreme disability) to 100 (no disability).
Change in Patient-specific functional scale (PSFS) | baseline and 12 weeks
  Patients will address one to three activities they have problems performing due to osteoarthritis. The degree of difficulty with performing these activities is rated from 0 (cannot perform the activity) to 10 (no problems).
Change in self-reported physical activity (International Physical Activity Questionnaire-Short Form) | baseline and 12 weeks
  Measured by The International Physical Activity Questionnaire-Short Form: Change in time (minutes per week/day) and Metabolic Equivalent of Task (MET-minutes per week/day) spent on sitting, walking, and moderate- and vigorous intensity physical activity the last week (0-7 days). METs are calculated by using the corresponding MET-values for walking (3.3 MET), and moderate-(4.0 MET) and vigorous (8.0 MET) intensity physical activity.
Change in self-reported physical activity (HUNT) | baseline and 12 weeks
  Measured by the three questions from the Nord-Trøndelag Health study (HUNT): change in average frequency (never/<1 per week/1 per week/2-3 per week/almost every day), intensity (easy without losing my breath or breaking into a sweat/so hard that I lose my breath and break into a sweat/I push myself to near-exhaustion) and duration (less than 15 minutes/15-29 minutes/30 minutes to 1 hour/more than 1 hour) of physical activity.
Change in self-reported pain intensity the last week | baseline and 12 weeks
  Measured by numeric rating scale ranging from 0 (no pain) to 10 (worst pain).
Change in self-reported fatigue the last week | baseline and 12 weeks
  Measured by numeric rating scale ranging from 0 (no fatigue) to 10 (worst fatigue).
Change in self-reported disease activity the last week | baseline and 12 weeks
  Measured by numeric rating scale ranging from 0 (good, no symptoms) to 10 (very bad, much symptoms).
Change in Health-related quality of life (EQ-5D-5L) | baseline and 12 weeks
  EQ-5D-5L will be used for measuring health-related quality of life (www.euroqol.org): comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels of answers (no problems, slight problems, moderate problems, severe problems, and extreme problems). The average score on each dimension will be reported, and the total score can be calculated into an index value ranging from -0.59 to 1, where -0.59 represents worst possible state and 1 represents perfect health.
Change in Arthritis Self-Efficacy Scale (ASES) | baseline and 12 weeks
  Measured by Arthritis Self-Efficacy Scale (ASES): comprises 11 items addressing pain and symptoms (scored on a 5-point scale ranging from not confident at all to very confident). The scores are summed up to a 0-100 score where higher score indicate better self-efficacy.
Change in exercise self-efficacy | baseline and 12 weeks
  Measured by Exercise Beliefs and Exercise Habits questionnaire: comprises 20 items addressing exercise self-efficacy (4 items), barriers to exercise (3 items), benefits of exercise (5 items), and impact of exercise on arthritis (8 items), scored on a 5-point Likert scale ranging from strongly disagree to strongly agree. The scores on each subscale is summed up where higher scores indicate better self-efficacy.

OTHER OUTCOMES:
Participant fidelity: proportion attending learning and mastery-course | baseline to 12 weeks
  Proportion of enrolled participants attending a 5-hour osteoarthritis learning and mastery-course (attendance registered by yes/no).
Participant fidelity (adherence): frequency of exercise | baseline to 12 weeks
  Total number of exercise sessions.
Participant fidelity (adherence): frequency of exercise per week | baseline to 12 weeks
  Average number of exercise sessions per week.
Participant fidelity (adherence): frequency of exercise weeks | baseline to 12 weeks
  Total number of weeks with minimum one exercise session.
Participant fidelity (adherence): duration of exercise sessions | baseline to 12 weeks
  Total number of exercise sessions completed according to prescribed duration. Measured by a question about completion of the prescribed exercise-session (yes/no).
Participant fidelity (adherence): intensity of exercise sessions | baseline to 12 weeks
  Total number of exercise sessions completed according to prescribed intensity. Measured by self-reported Rating of Perceived Exertion Scale (Borg RPE) ranging from 6 (resting) to 20 (maximal intensity).
Use of health care resources due to musculoskeletal pain | baseline
  Registered by self-report: 1) frequency (number of consultations the last 6 months) with a general practitioner and specialist health care (rheumatologist, orthopedist, neurologist, other), 2) referred (yes/no, the last 6 months) to x-ray, magnetic resonance imaging, physiotherapist, healthy life center, occupational therapist, 3) frequency (number of consultations during the last 6 months) with a physiotherapist, manual therapist, chiropractor, alternative treatment, other due, 4) had a stay at a rehabilitation institution during the last 6 months (yes/no and number of days). Descriptive data will be reported.
Use of medication due to musculoskeletal pain | baseline
  Registered by self-report: Frequency (never/<1 per month/monthly/weekly/daily/several times per day) of medication use (addressing pain, sleeping, depression, anxiety) the last 3 months will be self-reported through type, name and dosage (mg) of medication, in addition to use of other medication (yes/no) and type. Descriptive data will be reported.
Osteoarthritis pain on a Global Rating of Change scale | 12 weeks
  Change in osteoarthritis pain (from baseline to post-test) measured by a 7-point Global Rating of Change scale ranging from -3 (much worse) to +3 (much better).

CONTACTS AND LOCATIONS:
Overall Officials: Anne Therese Tveter, PhD, Principal Investigator — National Resource Center on Research in Rheumatology
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Data can possibly be made available on request

REFERENCES:
- [Derived] Joseph KL, Dagfinrud H, Hagen KB, Norden KR, Fongen C, Wold OM, Hinman RS, Nelligan RK, Bennell KL, Tveter AT. Adherence to a Web-based Exercise Programme: A Feasibility Study Among Patients with Hip or Knee Osteoarthritis. J Rehabil Med. 2023 Aug 14;55:jrm7139. doi: 10.2340/jrm.v55.7139. PMID 37578100
- [Derived] Joseph KL, Dagfinrud H, Hagen KB, Norden KR, Fongen C, Wold OM, Hinman RS, Nelligan RK, Bennell KL, Tveter AT. The AktiWeb study: feasibility of a web-based exercise program delivered by a patient organisation to patients with hip and/or knee osteoarthritis. Pilot Feasibility Stud. 2022 Jul 20;8(1):150. doi: 10.1186/s40814-022-01110-3. PMID 35859065